CLINICAL TRIAL: NCT02216370
Title: Detection of Occult Paroxysmal Atrial Fibrillation in Cryptogenic Stroke Patients or TIA Using an Implantable Loop Recorder and Correlation With Genetic Markers.
Brief Title: Detection of Occult Paroxysmal AF in Cryptogenic Stroke or TIA Patients Using an Implantable Loop Recorder and Correlation With Genetic Markers.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Martin (Other)
Responsible Party: Sponsor
Other Study IDs: NRRXT0001
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Cryptogenic Stroke or TIA; Atrial Fibrillation
Keywords: Cryptogenic stroke /TIA; Atrial Fibrillation; Implantable Loop Recorder; Genetic Mutation
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cryptogenic Stroke or TIA
- Healthy Volunteers: Healthy Volunteers as comparative group adjusted to investigated group by age and gender

SUMMARY:
Atrial fibrillation (AF) is the significant risk factor of ischemic stroke with incidence about 20% of all ischemic strokes. The undiagnosed AF in cryptogenic stroke patients could be present but not revealed by rutinne ECG.

DETAILED DESCRIPTION:
The subcutaneous Insertable Cardiac Monitor - Reveal® XT ICM, which provides long-term monitoring ( for 3 years), in selected stroke and TIA population on the basis of age, stroke etiology, and prescreening for cardiac arrhythmias helps to increase a detection of AF to 16.7% (range, 14.3% to 20.0%) in compare to ambulatory ECG detection of AF 6.4% (range, 5.3% to 9.0%). The AF detection after stroke and TIA strategically changes the therapeutic approach. In correlation with mentioned above the incidence of both specific genetic markers of AF and occurance of AF in this population and healthy volunteers are interesting.

ELIGIBILITY:
Inclusion Criteria:

* 1. Cryptogenic stroke or TIA within 72 h of onset symptoms according to the criteria for the Trial of Org 10172 in Acute Stroke Treatment (TOAST ) 2. National Institute of Health Stroke scale (NIHSS ) score ≤ 15 3. Modified Rankin Scale (mRS ) score ≤ 3 4. Ability and willingness of patients or their relatives or legal representatives to understand study instructions both verbal and written in accordance with ICH GCP and legislation applicable in the Slovak Republic

Exclusion Criteria:

* 1. Known etiology of stroke or TIA 2. Untreated hyperthyreosis 3. Myocardial infarct within 1 month of onset stroke or TIA 4. Coronary bypass within 1 month of onset stroke or TIA 5. Valvular disease requiring urgent surgery 6. Documented atrial fibrillation or flutter . 7. Patent Foramen Ovale (PFO) 8. Permanent indication to oral anticoagulation therapy 9. Long-term steroid therapy > 30 days 10. Participation in another clinical trial oriented to experimental pharmacologic therapy .

  11. Chronic inflammatory disease ( rheumatoid arthritide, IBD (Inflammatory bowel diseases ), lupus, vasculitis) 12. Severe co-morbidity not likely to complete to follow-up one year 13. Pregnant and breastfeeding women 14. Indication to pacemaker implantation, implantable cardioverter defibrillator (ICD) or Cardiac Resynchronization Therapy IPG or ICD implantation 15. Unabillity provide or unconsent with requiring protocol procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke or TIA confirmed by neurologist within 72 hours of onset symptoms
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Documented Atrial Fibrillation after episode of cryptogenic stroke / TIA Documented genetic mutation PITX2 and ZFHX3 | 12 months
  Documented Atrial Fibrillation after episode of cryptogenic stroke / TIA Documented genetic mutation PITX2 chromosome 4q25, polymorphism rs1906591,rs10033464 and ZFHX3 chromosome 16q22, polymorphism rs2106261

SECONDARY OUTCOMES:
Time to documented Atrial Fibrillation Reccurent stroke or TIA Stroke Secondary Prevention Therapy changes within 12 months Neuroimaging Changes ( brain CT/ MRI) | 12 months

OTHER OUTCOMES:
Follow-up of patients with implanted ECG monitor REVEAL XT incidence of atrial fibrillation, stroke or TIA | 3 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Nitra, Nitra, Slovakia

REFERENCES:
- [Derived] Petrovicova A, Kurca E, Brozman M, Hasilla J, Vahala P, Blasko P, Andrasova A, Hatala R, Urban L, Sivak S. Detection of occult paroxysmal atrial fibrilation by implantable long-term electrocardiographic monitoring in cryptogenic stroke and transient ischemic attack population: a study protocol for prospective matched cohort study. BMC Cardiovasc Disord. 2015 Dec 3;15:160. doi: 10.1186/s12872-015-0160-8. PMID 26631084